CLINICAL TRIAL: NCT01267500
Title: Randomized Study of Non-surgical Treatment Versus Observation in Asian Children With Intermittent Exotropia
Brief Title: Study of Non-surgical Treatment Versus Observation in Asian Children With Intermittent Exotropia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty to keep children in randomly assigned groups.
Sponsor: Singapore National Eye Centre (Other Government)
Responsible Party: Principal Investigator, Audrey Chia Wei-Lin, Senior Consultant, Singapore National Eye Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R765/49/2010
Record Dates: First submitted 2010-12-27; First posted 2010-12-28 (Estimated); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Intermittent Exotropia

ARMS (1):
- Non-surgical therapy (Experimental): patching or fusion exercises
  Interventions: Procedure: Non surgical therapy

INTERVENTIONS:
Procedure: Non surgical therapy — patching or fusion exercises

SUMMARY:
Non-surgical treatment (ie. patching or fusion exercises) of intermittent exotropia may help in increasing control of strabismus

ELIGIBILITY:
Inclusion Criteria:

1. Age 3 to 12 years (inclusive)
2. IXT for distance or constant IXT for distance and either IXT or exophoria for near
3. IXT size of > 10PD
4. Visual acuity in worse eye of at least 0.3 logMar (Snellen 6/12)
5. Visual acuity of no greater than 2 lines between eyes
6. Parents or guardian willing to accept randomization, and to continue with observation or treatment for at least 6-12 months, unless deterioration of strabismus or fall in best corrected visual acuity of worse than 0.3logMar (Snellen 6/12) in either eye
7. Investigator willing to observe IXT untreated for at least 1 year

Exclusion Criteria:

1. Previous non-surgical treatment for IXT, or patch treatment for amblyopia within the last year
2. Prior strabismus, intraocular or refractive surgery or botulinium injection
3. Surgery planned within the next year
4. Prematurity (birth weight < 1500g, gestational age < 34 weeks), systemic illness (eg. cerebral palsy), syndrome (including craniosynostosis) or learning disability
5. Any ocular abnormality (cornea, lens or central retina); nystagmus or conditions that limit eye movements.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Control of strabismus | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: audrey chia, Principal Investigator — Singapore National Eye Center
Locations (1):
- SIngapore National Eye Centre, Singapore, Singapore